CLINICAL TRIAL: NCT06193525
Title: FUnctional Selection of Advanced Breast Cancer Patients for Talazoparib Treatment Using the REpair Capacity (RECAP) Test: The FUTURE Trial
Brief Title: FUnctional Selection of Advanced Breast Cancer Patients for Talazoparib Treatment Using the REpair Capacity (RECAP) Test
Acronym: FUTURE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Leiden University Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dr. Agnes Jager MD, PhD, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 19-0070; 2018-002914-10 (EudraCT Number)
Record Dates: First submitted 2023-11-16; First posted 2024-01-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced Breast Cancer
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Talazoparib (Experimental): Talazoparib Capsule, oral use
  1 mg per day until PD or unacceptable toxicity
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Talazoparib is administered daily as single agent, 1 mg orally until unacceptable toxicity or progression of disease.
  Other Names: Talazoparib 1 MG Oral Capsule [Talzenna]

SUMMARY:
The goal of this clinical trial is to prove that the RECAP test is capable of selecting advanced breast cancer patients sensitive for treatment with the PARP inhibitor talazoparib. Participants will undergo an ultrasound-guided biopsy and a blood withdrawal. Homologous Recombination (HR) deficient patients (approximately 30%) can start talazoparib treatment until progression of the disease or unacceptable side-effects and their response will be evaluated.

DETAILED DESCRIPTION:
This is a single arm, prospective multicenter study among patients with advanced breast cancer with RECAP-based HRD phenotype who will be treated with talazoparib, a strong PARP inhibitor. After signing informed consent, metastatic breast cancer patients will undergo an ultrasound (or CT-) guided biopsy in order to obtain at least two biopsies from a metastatic lesion to determine the HR status by the RECAP test and a blood withdrawal for ctDNA isolation. HR proficient (HRP) patients will receive anti-tumor therapy (non study drug) on discretion of their treating physician; only the response on treatment will be registered. Approximately 30% of screened patients will have an HRD tumor and thus will be eligible to start talazoparib monotherapy until PD or unacceptable side effects. The primary endpoint is PFS at four months. Additional endpoints will include overall response rate and overall survival. Upon progression, patients will be kindly asked for consent to perform another biopsy (optional) and blood withdrawal in order to prove reversibility of the RECAP test outcome (from HRD to HRP) and explore potential mechanisms of resistance (both in tissue and ctDNA).

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status 0-2
* Locally advanced breast cancer without options for treatment with curative intent or metastatic breast cancer
* Objective progressive disease (PD) according to RECIST within 4 months prior to study entry
* The breast cancer must be either

  * high grade (Bloom & Richardson grade 3) ER positive (>10%) and HER2 negative primary breast cancer, or
  * triple negative (ER<10%, PR<10% and HER2 negative), or
  * any Bloom & Richardson grading and receptor status and also

    * at least one metastatic lesion must have a proven HRD phenotype based on a RECAP test not treated with anticancer therapy thereafter or
    * the patient must have a proven germline or somatic BRCA1 and/or BRCA2 mutation The Bloom & Richardson grading is always based on the primary tumor. The receptor status can be based on the primary tumor or a metastatic lesion whichever comes latest.
* The site of the metastatic lesion (or primary tumor in case it is still in situ) should be easily amendable for biopsy. NB lung metastases (high risk of hemato/pneumo-thorax) and bone metastases (not suitable for RECAP test because calcifications interfere with experimental procedures) are excluded. The local guidelines will be used for stopping and r estarting of anticoagulation. Bilirubin <1.5 ULN (except elevated bilirubin due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin) and both AST and ALT <5x ULN in case a liver biopsy is planned.
* The tumor must be HRD, defined as HRD identified by the RECAP test determined just before the start of potential Talazoparib treatment within this study (also in case a proven germline BRCA1/2 mutation is present).
* Maximum of four prior lines of chemotherapy for advanced disease; Patients who received platinum compounds are eligible if they have had at least a progression free interval of four months.
* Measurable or evaluable disease according to RECIST 1.1 criteria (appendix 2)
* Life expectancy ≥ 3 months
* Hemoglobin ≥ 10 g/dL (6,2 mmol/L) and ANC of ≥ 1.5 x 109 /L
* Platelets >100 x 10e9/L
* Hepatic function as defined by total serum bilirubin ≤ 1. 5 x ULN (except elevated bilirubin due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin), ASAT and ALAT < 3 x ULN or <5 x ULN in case of liver metastasis
* Adequate renal function as defined by either serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula)
* Negative pregnancy test (urine/serum) for female patients with childbearing potential
* Written informed consent

Exclusion Criteria:

* Any psychological condition potentially hampering compliance with the study protocol
* Any treatment with investigational antitumor drugs within 28 days prior to receiving the first dose of investigational treatment; or within 21 days for standard chemotherapy; or within 14 days for weekly scheduled chemotherapeutic regimens or endocrine therapy
* Radiotherapy within the last four weeks prior to receiving the first dose of investigational treatment; except 1 or 2 x 8 Gy for pain palliation, then seven days interval after the last radiation should be maintained
* Known persistent (>4 weeks) ≥ Grade 2 toxicity from prior cancer therapy (except for alopecia grade 2)
* Symptomatic brain or leptomeningeal metastases. Patients completely free of symptoms and without corticosteroids for at least four weeks after adequate treatment by resection and/or irradiation could be eligible (consult PI).
* Women who have a positive pregnancy test (urine/serum) and/or who are breastfeeding
* Unreliable contraceptive methods. Women and men enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: intra-uterine devices or systems, condom or other barrier contraceptive measures, sterilization and true abstinence)
* Concomitant use of P-gp inhibitors or inducers or BCRP inhibitors (see Appendix A)
* Any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Uncontrolled infectious disease (such as Human Immunodeficiency Virus HIV-1 or HIV-2 infection) or known active hepatitis B or C
* Recent myocardial infarction (< six months) or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with PFS at 4 months | Baseline. During the intervention: every 2 cycles (each cycle is 28 days), preferably within 7 days before the start of every uneven cycle. Follow-up until PD, unacceptable toxicity or death. Until all patients have reached PFS endpoint (end of study).
  The percentage of patients with advanced HRD breast cancer with PFS of 4 months or longer on talazoparib monotherapy. Disease assessment is performed by CT chest-abdomen per RECIST v 1.1.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Baseline. During the intervention: every 2 cycles (each cycle is 28 days), preferably within 7 days before the start of every uneven cycle. Follow-up until PD, unacceptable toxicity or death. Until all patients have reached PFS endpoint (end of study).
  The proportion of patients whose confirmed best overall response is either a PR or CR based upon investigator assessment per standard RECIST v1.1. Disease assessment is performed by CT chest-abdomen.
Overall survival (OS) | Time from first administration of talazoparib to time of death due to any cause. Follow-up on survival at least every 3 months for year 1, every 6 months for year 2 and 3 and annually until death. Until all patients have reached PFS (end of study).
  OS of patients with advanced HRD breast cancer treated with talazoparib

OTHER OUTCOMES:
Molecular aberrations in HR genes | A second biopsy at pre-screening
  Exploring differences in molecular aberrations in HR genes (e.g. BRCA1/2, PALB2). Based on between HRD tumors that respond and those that do not respond to talazoparib. Based on DNA analyses on snap-frozen biopsy taken at pre-screening.
PFS rate in relation to BRCA1/2 aberrations | A second biopsy at pre-screening
  PFS rate of non-BRCA1/2 or BRCA1 promoter methylated HRD tumors compared to PFS rate of BRCA1/2 mutated HRD tumors. Based on DNA analysis on snap-frozen biopsy taken at pre-screening.
Reversion of HRD phenotype | A second biopsy at pre-screening and optional: a biopsy at PD (immediately after the intervention). Until all patients have reached PFS endpoint (end of study).
  Exploring mechanisms of reversion of the HRD phenotype by comparing paired biopsies before treatment and upon progression on talazoparib.
Talazoparib resistance mechanisms in ctDNA | Blood samples will be taken at baseline and at PD (immediately after the intervention). Until all patients have reached PFS endpoint (end of study).
  Elucidating resistance mechanisms by sequencing a DNA repair gene panel on circulating tumor DNA (ctDNA) pretreatment and at disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Jager, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Groningen University Medical Center, Groningen